CLINICAL TRIAL: NCT05317013
Title: A Randomized, Double-Blind, Placebo-Controlled, Repeated-Dose Study to Assess the Safety, Tolerability, and Preliminary Effects of CHI-554 in Postmenopausal Women With Osteopenia
Brief Title: CBD in Postmenopausal Women With Osteopenia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: NM Clinical Research & Osteoporosis Center, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 710022US1314
Record Dates: First submitted 2022-03-21; First posted 2022-04-07 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - 100 mg CBD (Experimental): 100 mg CBD per day
  Interventions: Drug: CBD
- Group B - 300 mg CBD (Experimental): 300 mg CBD per day
  Interventions: Drug: CBD
- Group C - Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBD — CBD
  Arms: Group A - 100 mg CBD; Group B - 300 mg CBD
Other: Placebo — Placebo
  Arms: Group C - Placebo

SUMMARY:
This is a Phase 1, double-blind, placebo-controlled, repeated-dose study to assess the safety, tolerability, and preliminary effects of CHI-554 in postmenopausal women ages 50-80 years who have osteopenia.

ELIGIBILITY:
Inclusion Criteria:

* Is a female aged 50-80 years, inclusive, at the time of screening.
* Is postmenopausal, defined as > or = 12 months amenorrhoea.
* Has osteopenia, defined as T score at lumbar spine or femoral neck or total femur of less than -1.0, but not less than or equal to -2.5, according to dual energy x-ray absorptiometry (DXA) completed at the Screening Visit or performed at NM Clinical Research & Osteoporosis Center up to 6 months prior to the Screening Visit.
* Has been on a stable dose of 500 mg calcium daily for at least 7 days prior to Visit 1.
* Has a body mass index between 18 and 35 kg/m2 (inclusive).
* Is judged by the Investigator to be in generally good health at screening based on participants' medical history.
* Must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.

Exclusion Criteria:

* Has a history of epilepsy, hepatitis, or human immunodeficiency virus.
* Current or history of use of one or more prohibited medications (as described in Section 8.2.1.1).
* Changes in the use of a prescription, over-the-counter (OTC), systemic or topical drug(s), herbal supplement(s), or vitamin(s) for the 4 weeks prior to the Screening Visit.
* Evidence of clinically significant hepatic or renal impairment including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5× the upper limit of normal (ULN), or bilirubin >2× ULN.
* Has any clinically significant condition or abnormal finding at screening that would, in the opinion of the Investigator, preclude study participation or interfere with the evaluation of the study IP.
* Has a history of a known significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to cannabis, including phytocannabinoids and cannabinoid analogues, or excipients utilized within the IP (e.g., coconut; coconut oil; medium-chain triglycerides).
* Has taken grapefruit products and/or Seville oranges within the 7 days prior to Visit 1.
* Positive urine dipstick results for THC at the Screening Visit.
* Has a history or current diagnosis of a significant psychiatric disorder, including alcohol or substance use disorder, that would, in the opinion of the Investigator, affect the subject's ability to comply with the study requirements.
* Has participated in any investigational product or device study within 30 days prior to the Screening Visit, or is scheduled to participate in another investigational product or device study during the course of this study.
* Demonstrates behavior indicating unreliability or inability to comply with the requirements of the protocol.
* History of Osteoporosis diagnosis.

Ages: 50 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: Adverse Events/Serious Adverse Events | Week 4
  Adverse Events/Serious Adverse Events
Safety and Tolerability: Adverse Events/Serious Adverse Events | Week 8
  Adverse Events/Serious Adverse Events
Safety and Tolerability: Adverse Events/Serious Adverse Events | Week 12
  Adverse Events/Serious Adverse Events
Safety and Tolerability: Alanine aminotransferase (ALT) | Week 4
  Alanine aminotransferase
Safety and Tolerability: Alanine aminotransferase (ALT) | Week 12
  Alanine aminotransferase
Safety and Tolerability: Aspartate aminotransferase (AST) | Week 4
  Aspartate aminotransferase
Safety and Tolerability: Aspartate aminotransferase (AST) | Week 12
  Aspartate aminotransferase
Safety and Tolerability: Total bilirubin | Week 4
  Total bilirubin
Safety and Tolerability: Total bilirubin | Week 12
  Total bilirubin
Safety and Tolerability: Blood pressure | Week 4
  Blood pressure - Systolic and diastolic blood pressure
Safety and Tolerability: Blood pressure | Week 12
  Blood pressure - Systolic and diastolic blood pressure
Safety and Tolerability: Heart rate | Week 4
  Heart rate
Safety and Tolerability: Heart rate | Week 12
  Heart rate

SECONDARY OUTCOMES:
Serum CTx | Week 4
  Serum CTx
Serum CTx | Week 12
  Serum CTx
Serum P1NP | Week 4
  Serum P1NP
Serum P1NP | Week 12
  Serum P1NP
Serum Osteocalcin | Week 4
  Serum Osteocalcin
Serum Osteocalcin | Week 12
  Serum Osteocalcin
Serum Bone-specific alkaline phosphatase | Week 4
  Serum Bone-specific alkaline phosphatase
Serum Bone-specific alkaline phosphatase | Week 12
  Serum Bone-specific alkaline phosphatase

CONTACTS AND LOCATIONS:
Overall Officials: Lance Rudolph, MD, Principal Investigator — NM Clinical Research & Osteoporosis Center, Inc.
Locations (1):
- NM Clinical Research & Osteoporosis Center, Inc., Albuquerque, New Mexico, United States